CLINICAL TRIAL: NCT01936116
Title: Pain Perception and Side Effects During Sonohysterography With Balloon Catheters: a Randomized Comparative Study of Cervical With Uterine Catheter Placement
Brief Title: Optimal Balloon Catheter Placement During Sonohysterography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-Emb-016
Record Dates: First submitted 2013-08-25; First posted 2013-09-05 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2012-02

CONDITIONS: Infertility
Keywords: Sonohysterography; catheter placement; pain magnitude; vasovagal reaction
MeSH Terms: conditions — Infertility; Syncope, Vasovagal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients with intrauterine balloon catheter placement (Experimental): In this group, during the procedure of sonohysterography balloon catheter is inflated in the uterine cavity
  Interventions: Device: sonohysterography with inflated catheter in uterine cavity
- patients with intracervical balloon catheter placement (Active Comparator): During the procedure of sonohysterography balloon catheter is inflated in the cervical canal
  Interventions: Device: sonohysterography with inflated catheter in cervical cavity

INTERVENTIONS:
Device: sonohysterography with inflated catheter in uterine cavity — during the procedure of sonohysterography balloon catheter is inflated in the uterine cavity
  Arms: patients with intrauterine balloon catheter placement
Device: sonohysterography with inflated catheter in cervical cavity — During the procedure of sonohysterography balloon catheter is inflated in the cervical canal
  Arms: patients with intracervical balloon catheter placement

SUMMARY:
Saline infusion sonohysterography and other intrauterine investigations methods may cause uterine cramping, pain and vasovagal reactions. According to few of previous studies the position of catheter placement can affect the magnitude of pain and amount of saline required during the sonohysterography. The purpose of this double blind control trial study is to assess whether the location of the balloon catheter either the uterus or cervix during sonohysterography can affect the magnitude of pain and the rate of vasovagal reaction.

DETAILED DESCRIPTION:
The proposal of study approved by the investigators institutional review boards and institution's ethical committee, and all participants will sign a written consent before enter to study. A total of 300 infertile women undergoing sonohysterography will be randomized to intrauterine or intracervical balloon catheter placement. The examination is scheduled in the early follicular phase of menstrual cycle, immediately after cessation of menstrual flow and before day 10. After preparation of patient, a 2 lumen 6-French flexible catheter is introduced into the cervical canal and balloon at the catheter tip is placed in the lower uterine segment or 1 cm into cervical canal and inflated with 1 mL of sterile saline solution. Under sonographic guidance, sterile normal saline solution (10-50 mL) is slowly introduced into the cavity until an adequate distention of the uterine cavity is obtained. Three-dimensional ultrasound scanned volumes are recorded. Patients are asked to assess their level of pain at the time of the balloon inflation and deflation using a 10-point visual analog pain scale. Patients are checked for the sign and symptoms of vasovagal reaction during and 30 minutes after procedure. Outcome measures will be assessed based on the intent-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients who will be referred to Royan institute for sonohysterography to evaluate the internal structure of uterine cavity (acquired & congenital abnormalities) are included in this prospective comparative study.

Exclusion Criteria:

* Exclusion Criteria:

  * Symptoms of active pelvic infection
  * Abnormal uterine bleeding
  * Women with cervical stenosis
  * Women with each lesions which disrupts catheterization such as large myoma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
perceived Pain | during sonohysterography
  inflation of the balloon & deflation of the balloon by a 10-point visual analog pain scale
Vasovagal reactions | During sonohysterography
  Evaluation the vasovagal reactions (Hypotension, vomiting, syncope)in patients During procedure .
vasovagal reaction | 30 minutes after sonohysterography
  Evaluation the vasovagal reactions (Hypotension, vomiting, syncope)in patients 30 minutes after procedure .

SECONDARY OUTCOMES:
Saline volume | during sonohysterography
  Evaluation the saline volume that is required for sonohisterography
time of procedure | during sonohysterography
  Evaluation the total time that is needed for sonohysterography.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Fatemeh Zafarani, MSc, Study Director — Department of Reproductive Imaging at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine; Firoozeh Ahmadi, MD, Principal Investigator — Department of Reproductive Imaging at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.org